CLINICAL TRIAL: NCT02188160
Title: A Phase II, Double-Masked, Randomized, Controlled Study of KPI-121 0.25% Ophthalmic Suspension Compared to Vehicle in Subjects With Dry Eye Disease
Brief Title: Safety and Efficacy of KPI-121 in Subjects With Dry Eye Disease
Acronym: Kauai
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Kala Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: KPI-121-C-002
Record Dates: First submitted 2014-07-09; First posted 2014-07-11 (Estimated); Results first posted 2021-01-06 (Actual); Last update posted 2021-01-06 (Actual); Status verified 2019-07

CONDITIONS: Dry Eye Syndromes; Keratoconjunctivitis Sicca
Keywords: Pain; Corticosteroid; Dry Eye; Hyperemia; Ocular Discomfort
MeSH Terms: conditions — Dry Eye Syndromes; Keratoconjunctivitis Sicca; Pain; Hyperemia | interventions — Loteprednol Etabonate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- KPI-121 0.25% Ophthalmic Suspension (Active Comparator): KPI-121 0.25% ophthalmic suspension dosed QID for 28 days in subjects with dry eye disease
  Interventions: Drug: KPI-121
- Vehicle (Placebo Comparator): Vehicle (placebo) dosed QID for 28 days in subjects with dry eye disease
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: KPI-121 — KPI-121 drug product will be supplied as 0.25% as a suspension in identically packaged opaque dropper bottles. KPI-121 drug product is a sterile, aqueous, submicron suspension of loteprednol etabonate.
  Other Names: KPI-121 0.25% Ophthalmic Suspension; Loteprednol etabonate
  Arms: KPI-121 0.25% Ophthalmic Suspension
Drug: Placebo — Subjects randomized to placebo control arms will receive the same bottles containing all components at the concentrations used in the KPI-121 drug product with the exception of the active component, loteprednol etabonate.
  Other Names: Vehicle of KPI-121 0.25% Ophthalmic Suspension
  Arms: Vehicle

SUMMARY:
The primary purpose of this study is to determine the efficacy and safety of KPI-121 0.25% ophthalmic suspension compared to vehicle (placebo) in subjects who have a documented clinical diagnosis of dry eye disease. The product will be studied over 28 days, with 1-2 drops instilled in each eye four times daily (QID).

DETAILED DESCRIPTION:
This is a Phase II, multi-center, double-masked, randomized, vehicle-controlled, parallel-group study designed to evaluate the safety and efficacy of KPI-121 0.25% ophthalmic suspension versus vehicle in subjects with dry eye disease.

Approximately 400 subjects will be screened and up to 150 subjects will be randomized at up to 12 centers located in the United States. Subjects will be randomized to 1 of 2 study arms in an approximate 1:1 ratio. The study arms are: 1) KPI-121 0.25% ophthalmic suspension administered 1-2 drops in each eye QID for up to 28 days or 2) vehicle administered as 1-2 drops in each eye QID for up to 28 days.

This study will include up to 6 clinic visits over 6 weeks. At Visit 1 Screening (14 ± 1 days prior to Day 1), subjects who meet screening inclusion/exclusion criteria will begin a 2-week run-in period during which they will be treated with 1-2 drops of single-masked vehicle in each eye QID for 14 ± 1 days.

At Visit 2, Randomization (Day 1), subjects who continue to meet inclusion/exclusion criteria will be eligible for randomization to 1 of the 2 arms of the study (i.e., KPI-121 0.25% ophthalmic suspension or vehicle). Following randomization, subjects will be instructed to return to the clinic to have a complete study evaluation at Study Visits 4 and 6 (Days 15 ± 1 day and 29 ± 1 day, respectively). Subjects will further be instructed to return to the clinic for diary collection and in-clinic symptom assessment only at Visits 3 and 5 (Days 8 ± 1 day and 22 ± 1 day, respectively). The last dose of investigational product and the final study visit will occur upon completion of 28 ± 1 days of exposure to investigational product. Subjects will be released from the study at the end of Visit 6 (Day 29 ± 1 day).

ELIGIBILITY:
Inclusion Criteria:

• Have a documented clinical diagnosis of dry eye disease in both eyes

Exclusion Criteria:

* Known hypersensitivity/contraindication to study product(s) or components.
* History of glaucoma, IOP >21 mmHg at the screening or randomization visits, or being treated for glaucoma in either eye.
* Diagnosis of: ongoing ocular infection; severe/serious ocular condition that in judgment of Investigator could confound study assessments or limit compliance; severe/serious systemic disease or uncontrolled medical condition that in judgment of Investigator could confound study assessments or limit compliance; or have been exposed to an investigational drug within the 30 days prior to screening.
* In the opinion of Investigator or study coordinator, be unwilling or unable to comply with study protocol or unable to successfully instill eye drops.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2014-06; Primary Completion 2015-01 (Actual); Study Completion 2015-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gregg Berdy, MD, Principal Investigator — Ophthalmology Associates; David Evans, OD, Principal Investigator — Total Eye Care, PA; Kathy Kelley, OD, Principal Investigator — Price Vision Group; Joseph Martel, MD, Principal Investigator — Martel Eye Medical Group; Mark Milner, MD, Principal Investigator — Eye Center of Southern CT, P.C.; Steven Rauchman, MD, Principal Investigator — North Valley Eye Medical Group; Kenneth Sall, MD, Principal Investigator — Sall Research Medical Center; Jeffrey Whitsett, MD, Principal Investigator — Whitsett Vision Group; Marc Abrams, MD, Principal Investigator — Abrams Eye Center; Michael Korenfeld, MD, Principal Investigator — Ecomprehensive Eye Care, Ltd / Vision Research Institute LLC; Jodi Luchs, MD, Principal Investigator — South Shore Eye Center
Locations (11):
- United States (11):
  - Sall Research Medical Center, Artesia, California
  - North Valley Eye Medical Group, Mission Hills, California
  - Martel Eye Medical Group, Rancho Cordova, California
  - Eye Center of Southern CT, P.C., Hamden, Connecticut
  - Price Vision Group, Indianapolis, Indiana
  - Ophthalmology Associates, St Louis, Missouri
  - Comprehensive Eye Care, Ltd. / Vision Research Institute, LLC, Washington, Missouri
  - South Shore Eye Center, LLP, Wantagh, New York
  - Abrams Eye Center, Cleveland, Ohio
  - Total Eye Care, PA, Memphis, Tennessee
  - Whitsett Vision Group, Houston, Texas

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Korenfeld M, Nichols KK, Goldberg D, Evans D, Sall K, Foulks G, Coultas S, Brazzell K. Safety of KPI-121 Ophthalmic Suspension 0.25% in Patients With Dry Eye Disease: A Pooled Analysis of 4 Multicenter, Randomized, Vehicle-Controlled Studies. Cornea. 2021 May 1;40(5):564-570. doi: 10.1097/ICO.0000000000002452. PMID 32826644

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | KPI-121 0.25% Ophthalmic Suspension | Vehicle
Started | 73 | 77
Completed | 72 | 76
Not Completed | 1 | 1
Not completed — Adverse Event | 1 | 0
Not completed — Use of an excluded medication | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | KPI-121 0.25% Ophthalmic Suspension | Vehicle | Total
Number analyzed (Participants) | 73 | 77 | 150
Age, Continuous [Mean (Standard Deviation); unit: years] | 56.3 (17.17) | 54.9 (12.29) | 55.6 (14.83)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 53 | 61 | 114
  Male | 20 | 16 | 36
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 15 | 16 | 31
  Not Hispanic or Latino | 58 | 61 | 119
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 3 | 4 | 7
  Native Hawaiian or Other Pacific Islander | 2 | 1 | 3
  Black or African American | 10 | 8 | 18
  White | 54 | 63 | 117
  More than one race | 0 | 1 | 1
  Unknown or Not Reported | 4 | 0 | 4
Region of Enrollment [Number; unit: participants]
  United States | 73 | 77 | 150

OUTCOME MEASURES:

1. Primary Outcome: Bulbar Conjunctival Hyperemia
Description: Comparison of mean bulbar conjunctival hyperemia in the study eye between the KPI-121 0.25% ophthalmic suspension group and the vehicle group using a 0-4 grading scale. The grading scale was based on the Cornea and Contact Lens Research Unit Grading Scale where 0 = none, 1 = very slight, 2 = slight, 3 = moderate and 4 = severe.
Time Frame: Visit 6 (Day 29)
Population: ITT
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | KPI-121 0.25% Ophthalmic Suspension | Vehicle
Number analyzed (Participants) | 73 | 77
score on a scale | 1.22 (0.633) | 1.36 (0.626)

2. Primary Outcome: Ocular Discomfort
Description: Comparison of mean ocular discomfort severity between the KPI-121 0.25% ophthalmic suspension group and the vehicle group using a 0-100 visual analog grading scale where 0 was better and 100 was worse.
Time Frame: Visit 6 (Day 29)
Population: ITT
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | KPI-121 0.25% Ophthalmic Suspension | Vehicle
Number analyzed (Participants) | 73 | 77
score on a scale | 57.05 (23.892) | 60.47 (19.770)

3. Secondary Outcome: Corneal Fluorescein Staining Scores
Description: Comparison of mean corneal fluorescein staining scores in the study eye between the KPI-121 0.25% ophthalmic suspension group and the vehicle group using methods developed by the National Eye Institute (NEI) Dry Eye Workshop in evaluating 5 regions of the cornea (superior, inferior, nasal, temporal and central) using a 0-3 grading scale, where 0 = no visible staining, 1 = Mild, 2 = moderate and 3 = severe. The total score is obtained by summing each of the 5 sections of the cornea. The NEI score will be from 0-15.
Time Frame: Visit 4 (Day 15) and Visit 6 (Day 29)
Population: ITT
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | KPI-121 0.25% Ophthalmic Suspension | Vehicle
Number analyzed (Participants) | 73 | 77
score on a scale
  Visit 4 (Day 15) | 6.15 (2.582) | 7.00 (2.920)
  Visit 6 (Day 29) | 5.64 (2.889) | 6.16 (3.445)

4. Secondary Outcome: Bulbar Conjunctival Hyperemia Scores
Description: Comparison of mean bulbar conjunctival hyperemia scores in the study eye between the KPI-121 0.25% ophthalmic suspension group and the vehicle group using a 0-4 grading scale. The grading scale was based on the Cornea and Contact Lens Research Unit Grading Scale where 0 = none, 1 = very slight, 2 = slight, 3 = moderate and 4 = severe.
Time Frame: Visit 4 (Day 15)
Population: ITT
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | KPI-121 0.25% Ophthalmic Suspension | Vehicle
Number analyzed (Participants) | 73 | 77
score on a scale | 1.36 (0.586) | 1.42 (0.676)

5. Secondary Outcome: Ocular Discomfort
Description: as for outcome 2
Time Frame: Visit 4 (Day 15)
Population: ITT
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | KPI-121 0.25% Ophthalmic Suspension | Vehicle
Number analyzed (Participants) | 73 | 77
score on a scale | 58.83 (20.745) | 63.63 (17.844)

ADVERSE EVENTS:
Time Frame: Adverse event data was collected from Visit 2 (Day 1) through Visit 6 (Day 29).
Description: One Subject was randomized to KPI-121 0.25% but received vehicle. Therefore, 72 subjects are included in the KPI-121 0.25% group and 78 subjects are included in the vehicle group in the safety analyses.
Arm/Group | KPI-121 0.25% Ophthalmic Suspension | Vehicle
All-Cause Mortality (participants affected / at risk) | 0/72 | 0/78
Serious Adverse Events (participants affected / at risk) | 1/72 | 0/78
Other Adverse Events (participants affected / at risk) | 7/72 | 8/78
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | KPI-121 0.25% Ophthalmic Suspension (N=72) | Vehicle (N=78)
Cholelithiasis (Hepatobiliary disorders) | 1 (1) | 0 (0) — One subject reported an SAE (cholelithiasis; KPI-121 0.25% group), which was considered unrelated to the study treatment; it was severe in intensity, led the subject to discontinue the study treatment, and ultimately resolved without sequelae.
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | KPI-121 0.25% Ophthalmic Suspension (N=72) | Vehicle (N=78)
Instillation site pain (General disorders) | 7 (18) | 8 (16)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The institution and Investigators participating in this trial shall have no right to publish or present the results of this study without the prior written consent of the sponsor.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2014-09-26): https://cdn.clinicaltrials.gov/large-docs/60/NCT02188160/Prot_SAP_000.pdf